CLINICAL TRIAL: NCT03818178
Title: Intramyocellular Fatty Acid Trafficking in Insulin Resistance States - Effects of Intestinal Delivery of Lipids
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michael D. Jensen, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18-002520; 5R01DK045343-27 (NIH)
Record Dates: First submitted 2019-01-20; First posted 2019-01-28 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — soybean oil, phospholipid emulsion; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intralipid (Experimental)
  Interventions: Dietary Supplement: Intralipid
- Palm Oil (Experimental)
  Interventions: Dietary Supplement: Palm Oil Emulsion
- Saline (Placebo Comparator)
  Interventions: Other: Saline

INTERVENTIONS:
Dietary Supplement: Intralipid — Half of the participants will receive either naso-duodenal infusion of intralipid or palm oil each participant will serve as their own saline control on the second study day.
  Arms: Intralipid
Dietary Supplement: Palm Oil Emulsion — Half of the participants will receive either naso-duodenal infusion of intralipid or palm oil each participant will serve as their own saline control on the second study day.
  Arms: Palm Oil
Other: Saline — All participants will serve as their own controls with a saline infusion study day.
  Arms: Saline

SUMMARY:
Muscle insulin resistance is a hallmark of upper body obesity (UBO) and Type 2 diabetes (T2DM). It is unknown whether muscle free fatty acid (FFA) availability or intramyocellular fatty acid trafficking is responsible for muscle insulin resistance, although it has been shown that raising FFA with Intralipid can cause muscle insulin resistance within 4 hours. The investigators do not understand to what extent the incorporation of FFA into ceramides or diacylglycerols (DG) affect insulin signaling and muscle glucose uptake. The investigators propose to alter the profile and concentrations of FFA of healthy, non-obese adults using an overnight, intra-duodenal palm oil infusion vs. an overnight intra-duodenal Intralipid infusion (both compared to saline control). The investigators will compare the muscle FFA storage into intramyocellular triglyceride, intramyocellular fatty acid trafficking, activation of the insulin signaling pathway and glucose disposal rates, providing the first measure of how different FFA profiles alter muscle FFA trafficking and insulin action at the whole body and cellular/molecular levels. By identifying which steps in the insulin signaling pathway are most affected, the investigators will determine the site-specific effect of ceramides and/or DG on different degrees of insulin resistance.

Hypothesis 1: Palm oil infusion will result in abnormal FFA trafficking into intra-myocellular ceramides and abnormal insulin signaling.

Hypothesis 2: Intralipid infusion will result in abnormal FFA trafficking into intra-myocellular saturated DG and abnormal insulin signaling.

ELIGIBILITY:
Inclusion Criteria:

* Women and Men (Women premenopausal)
* BMI 18-27
* Weight stable
* Not pregnant/nursing

Exclusion Criteria:

* Ischemic heart disease
* Atherosclerotic valvular disease
* Smokers (> 20 cigarettes per week)
* Bilateral oophorectomy
* Concomitant use of medications that can alter serum lipid profile (high dose fish oil, statins, niacin, fibrates, thiazolinediones, beta-blockers, atypical antipsychotics)
* Lidocaine allergy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in fatty acid enrichment of intramyocellular signaling molecules before and after a euglycemic, hyperinsulinemic clamp | 18 hours
  The study involves the use of a hyperinsulinemic, euglycemic clamp to compare fatty acid enrichments in intramyocellular signaling molecules. The first half of the study will be the "pre-clamp" stage. During this stage, volunteers will receive an intravenous infusion of C13-labelled palmitate as a tracer in order for enrichment calculations to be performed pre-clamp. One muscle biopsy will be obtained to measure fatty acid enrichment within intramyocellular ceramides, diacylglycerols, long-chain acylcarnitines, and intramyocellular triglycerides. The insulin clamp will then commence, and volunteers will simultaneously receive an intravenous infusion of a second tracer, D-9 palmitate. This tracer will allow us to calculate enrichments during the insulin clamp stage of the study. A second muscle biopsy will be performed at the end of the insulin clamp, and similar enrichment calculations will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Jensen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials